CLINICAL TRIAL: NCT00074074
Title: Randomized Phase II Trial With Infliximab (Remicade) in Patients With Myelodysplastic Syndrome and a Relatively Low Risk of Developing Acute Leukemia
Brief Title: Infliximab in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-06023; EORTC-06023
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory | interventions — Infliximab

INTERVENTIONS:
Biological: infliximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as infliximab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Randomized phase II trial to study the effectiveness of infliximab in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic activity of 2 different doses of infliximab on peripheral blood cell count and peripheral and bone marrow blast cell count in patients with low- or intermediate-risk myelodysplastic syndromes.
* Determine the subjective and objective toxicity of these regimens in these patients.
* Determine the response rates (complete and partial response and hematological improvement) in patients treated with these regimens.
* Determine the duration of response in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to cytogenetics (good vs intermediate vs unknown due to failure), overall International Prognostic Scoring System score (low [0] vs intermediate 1 [0.5-1.0] vs intermediate 2 [1.5-2.0]), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive infliximab IV on days 1, 15, 43, 71, 99, 127, 155, and 183 in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive a higher dose of infliximab as in arm I. Patients achieving response (complete or partial response or hematological improvement) continue therapy beyond day 183 in the absence of disease progression.

Patients are followed at 2 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 80 patients (40 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis (within the past month) of low- or intermediate-risk myelodysplastic syndromes (MDS) meeting all of the following criteria:

  * No more than 10% bone marrow blasts (corresponding to refractory anemia [RA], RA with ringed sideroblasts, or RA with excess blasts)
  * Meets at least 1 of the following hematopoietic criteria:

    * Hemoglobin no greater than 10 g/dL OR red blood cell transfusion dependent
    * Neutrophil count no greater than 1,500/mm^3
    * Platelet count no greater than 100,000/mm^3 OR platelet transfusion dependent
  * No poor cytogenetics (complex abnormalities or involvement of chromosome 7)

    * Patients with unknown cytogenetics may be eligible provided reasonable efforts have been made for determining the cytogenetic profile and the results are considered a failure (e.g., normal karyotype [NN] with no more than 10 metaphases)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* No history of documented hepatitis C
* No documented active hepatitis B
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT less than 2.5 times ULN

Renal

* Creatinine less than 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease
* No clinical history or evidence of congestive heart failure
* No severe cardiac dysfunction
* LVEF greater than 35%

Pulmonary

* No prior or concurrent active or latent tuberculosis (TB)

  * No evidence of prior or concurrent active TB (i.e., fibrotic or pleural scarring, pulmonary nodules, mediastinal and/or hilar lymphadenopathy, upper lobe volume loss, or cavitation) by chest x-ray
  * Negative intradermal tuberculin skin test (i.e., induration less than 5 mm)
* No severe pulmonary dysfunction

Immunologic

* No prior or concurrent opportunistic infection (e.g., herpes zoster, cytomegalovirus, Pneumocystic carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within the past 6 months
* No concurrent severe (CTC grade III or IV) active, chronic, or recurrent infections
* No recent history of allergies
* HIV negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No prior clinically significant adverse event to murine or chimeric proteins or human/murine recombinant products
* No recent contact with an individual with active TB
* No poor medical risk due to other systemic disease
* No multiple sclerosis or other demyelinating disorder
* No peripheral neuropathy greater than CTC grade 1
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior infliximab or other monoclonal antibodies
* At least 6 weeks since prior hematopoietic growth factors for MDS
* At least 3 months since prior therapy targeted at reducing tumor necrosis factor (TNF) alpha (e.g., pentoxifylline, thalidomide, or etanercept)
* No concurrent epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF)
* No other concurrent drugs targeted at reducing TNF alpha (e.g., pentoxifylline, thalidomide, or etanercept)

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior solid organ transplantation

  * Corneal transplantation more than 3 months ago allowed

Other

* No prior randomization to this clinical trial
* At least 6 weeks since prior treatment for MDS (except supportive care)
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent therapeutic-dose nonsteroidal anti-inflammatory drugs (NSAIDs)

  * Concurrent sporadic (no more than 3 tablets/week) over-the-counter NSAIDs allowed
* Concurrent cardioprotective doses (80 mg/day or equivalent) of aspirin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-10; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Best response as measured by Cheson response criteria

SECONDARY OUTCOMES:
Duration of highest grade toxicity as assessed by CTCAE v3.0 after response

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Zwierzina, MD, Study Chair — Medical University Innsbruck
Locations (19):
- Belgium (7):
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - H. Hartziekenhuis - Roeselaere., Roeselare
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- Czechia (2):
  - University Hospital - Olomouc, Olomouc
  - Institute of Hematology and Blood Transfusion, Prague
- France (2):
  - Centre Antoine Lacassagne, Nice
  - Hotel Dieu de Paris, Paris
- Germany (3):
  - Ruprecht - Karls - Universitaet Heidelberg, Heidelberg
  - Marienhospital Stuttgart, Stuttgart
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
- Ospedale San Salvatore, Pesaro, Italy
- Netherlands (4):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Ziekenhuis Bronovo, The Hague

REFERENCES:
- [Result] Baron F, Suciu S, Amadori S, Muus P, Zwierzina H, Denzlinger C, Delforge M, Thyss A, Selleslag D, Indrak K, Ossenkoppele G, de Witte T. Value of infliximab (Remicade(R)) in patients with low-risk myelodysplastic syndrome: final results of a randomized phase II trial (EORTC trial 06023) of the EORTC Leukemia Group. Haematologica. 2012 Apr;97(4):529-33. doi: 10.3324/haematol.2011.044347. Epub 2011 Nov 18. PMID 22102701
- [Result] Baila L, Suciu S, Muus P, et al.: Assessment of two doses of infliximab in patients with low/intermediate risk IPSS myelodysplastic syndrome (MDS): an EORTC leukemia group (LG) randomized phase II trial (06023). [Abstract] Blood 110 (11): A-1456, 2007.